CLINICAL TRIAL: NCT06851117
Title: Compare The Effectiveness of Spider Cage Therapy and Proprioceptive Neuromuscular Facilitation (PNF) In Children With Cerebral Palsy
Brief Title: Compare The Effectiveness of SCT and PNF In Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/754
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Neuromuscular Facilitation (PNF) (Experimental)
  Interventions: Combination Product: Proprioceptive Neuromuscular Facilitation (PNF)
- Spider Cage Therapy Group (Experimental)
  Interventions: Combination Product: Spider Cage Therapy Group
- Combined PNF and Spider Cage Therapy Group (Active Comparator)
  Interventions: Diagnostic Test: Combined PNF and Spider Cage Therapy Group

INTERVENTIONS:
Combination Product: Proprioceptive Neuromuscular Facilitation (PNF) — Participants in the PNF group will undergo intensive training of the affected limbs for 20 minutes per day, 5 days a week, over a 4-week period. During therapy sessions, the unaffected limb will be constrained using a mitt or cast to encourage focused activation and strengthening of the affected side. The therapy will include repetitive movement patterns designed to enhance strength, flexibility, and coordination.
  Arms: Proprioceptive Neuromuscular Facilitation (PNF)
Combination Product: Spider Cage Therapy Group — This group will participate in therapy sessions within the Spider Cage for 20 minutes per day, 5 days a week, for 4 weeks. Interventions will involve weight-bearing exercises, movement facilitation, and balance training, utilizing the cage's elastic cords to support and stabilize posture. The goal is to improve gross motor skills, balance, and controlled movement.
  Arms: Spider Cage Therapy Group
Diagnostic Test: Combined PNF and Spider Cage Therapy Group — Participants in this group will receive both PNF and Spider Cage Therapy, with integrated principles and techniques from both approaches. The intensity and duration will be consistent with the individual therapy groups, with sessions held for 20 minutes per day, 5 days a week, over 4 weeks. This combination is expected to enhance functional outcomes by targeting both strength/coordination and balance/postural control.
  Arms: Combined PNF and Spider Cage Therapy Group

SUMMARY:
This study will evaluate the comparative effectiveness of Spider Cage Therapy (SCT) and Proprioceptive Neuromuscular Facilitation (PNF) in managing motor impairments in children with cerebral palsy (CP). Cerebral palsy often leads to motor deficits that limit movement and impair functionality.

DETAILED DESCRIPTION:
SCT and PNF are therapeutic interventions that target these motor challenges but use distinct approaches. Spider Cage Therapy will involve the use of elastic cords within a supportive frame (the "spider cage") to stabilize the child, enhancing postural control and enabling dynamic movement training. This approach is expected to improve balance and alignment, promoting functional mobility. In contrast, PNF will focus on neuromuscular reeducation through specific movement patterns intended to enhance strength, coordination, and flexibility. By comparing SCT and PNF, this study aims to identify their respective impacts on motor function improvements, particularly in gross motor skills, balance, and postural stability, potentially guiding future rehabilitation protocols for children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-12 years.
* Clinical diagnosis of cerebral palsy.
* Classified within Gross Motor Function Classification System (GMFCS) levels I to III.
* Ability to follow instructions and participate in therapy sessions.

Exclusion Criteria:

* Severe cognitive impairments hindering participation.
* Severe musculoskeletal deformities or recent surgeries.
* Other medical conditions contraindicating participation in physical therapy.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-66 | 12 Months
  Five levels and each has different nbr of questions each having 0- 3 score 0 no movement 3 complete movement
Paedetric balance scale | 12 months
  14 items each have 0-4 score total 56 0 totally dependent 4 independently can prrform movement
Functional Independence Measure for Children (WeeFIM) | 12 months
  for overall functional independence (FIM) it has total 18 items 13 relatesd to mobilty and 5 regarding cognition Each has1- 7 score where reports total dependence and 7 shows complete independence

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No